CLINICAL TRIAL: NCT05927350
Title: Research Participation With Transgender and Gender-Diverse Youth
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: HM20026635
Record Dates: First submitted 2023-06-02; First posted 2023-07-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Transgender Persons
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Survey: Participants will complete a one-time survey asking about sociodemographics, pediatric research participation, experience with research, gender minority stress and resilience, vaccine hesitancy, medical mistrust, and connectedness to the LGBT community
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey asking about sociodemographics, pediatric research participation, experience with research, gender minority stress and resilience, vaccine hesitancy, medical mistrust, and connectedness to the LGBT community

SUMMARY:
Research has historically excluded the participation of transgender and gender-diverse people. The purpose of this research study is to find out about what goes into a transgender and gender-diverse youth's decision to participate in research. The results of this study will be used to improve access to research for transgender and gender-diverse youth and therefore, improve the representation of transgender and gender-diverse youth as research participants in research.

ELIGIBILITY:
Inclusion Criteria:

* Gender identity different then sex assigned at birth
* Between the ages 15-21 years

Exclusion Criteria:

* Gender identity the same as their sex assigned at birth
* Younger than 15 years of age, and older than 21 years of age

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Gender identity different then sex assigned at birth and ages 15-21 years
Study Population: Transgender and gender-diverse adolescents
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quantitative Assessment of Pediatric Research Participation in Transgender Youth | through study completion, estimated to be 3 months
  The outcome will be the responses (agree or disagree) to the different items in the Pediatric Research Participation measure.
Qualitative Assessment of Pediatric Research Participation in Transgender Youth | through study completion, estimated to be 3 months
  The investigators will implement qualitative analysis to explore transgender and gender-diverse youths experiences with research, and barriers and facilitators to participating in research. Specifically, the outcomes will be themes and supporting quotes.

CONTACTS AND LOCATIONS:
Overall Officials: An Pham, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No